CLINICAL TRIAL: NCT01670877
Title: A Phase II Study of Neratinib Alone and in Combination With Fulvestrant in Metastatic HER2 Non-amplified But HER2 Mutant Breast Cancer
Brief Title: Neratinib +/- Fulvestrant in Metastatic HER2 Non-amplified But HER2 Mutant Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Puma Biotechnology, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201209135
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Breast Neoplasms
Keywords: Neratinib; fulvestrant; HER2 mutation; metastatic breast cancer; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Fulvestrant; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part I: Neratinib Only (Experimental): -Patients will receive neratinib PO daily on Days 1-28. Each cycle is 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Neratinib; Procedure: Tumor biopsy; Procedure: Research blood sample
- Part II: Neratinib Only (ER-) (Experimental): -Patients will receive neratinib PO daily on Days 1-28. Each cycle is 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Neratinib; Procedure: Tumor biopsy; Procedure: Research blood sample
- Part II: Neratinib + Fulvestrant (ER+, fulvestrant-naive) (Experimental): -Patients will receive neratinib PO daily on Days 1-28 and fulvestrant on Day 1 of each cycle (and C1D15). Each cycle is 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Neratinib; Drug: Fulvestrant; Procedure: Tumor biopsy; Procedure: Research blood sample
- Part II: Neratinib + Fulvestrant (ER+. prior fulvestrant-tx) (Experimental): -Patients will receive neratinib PO daily on Days 1-28 and fulvestrant on Day 1 of each cycle (and C1D15). Each cycle is 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Neratinib; Drug: Fulvestrant; Procedure: Tumor biopsy; Procedure: Research blood sample
- Crossover: Neratinib + Trastuzumab (Experimental): -If a participant experiences disease progression during Part I or Part II following neratinib, trastuzumab (or FDA approved biosimilar) may be added to the treatment regimen. Trastuzumab may be administered intravenously with a loading dose of 6 mg/kg then 4 mg/kg every 2 weeks. A cycle will be defined as 28 days. Patients will continue to receive neratinib PO daily on Days 1-28. Each cycle is 4 weeks.
  Interventions: Drug: Neratinib; Drug: Trastuzumab; Procedure: Tumor biopsy; Procedure: Research blood sample
- Crossover: Neratinib + Fulvestrant + Trastuzumab (Experimental): -If a participant experiences disease progression during Part I or Part II following neratinib, trastuzumab (or FDA approved biosimilar) may be added to the treatment regimen. Trastuzumab may be administered intravenously with a loading dose of 6 mg/kg then 4 mg/kg every 2 weeks. A cycle will be defined as 28 days. Patients will receive neratinib PO daily on Days 1-28 and fulvestrant on Day 1 of each cycle (and C1D15). Each cycle is 4 weeks.
  Interventions: Drug: Neratinib; Drug: Fulvestrant; Drug: Trastuzumab; Procedure: Tumor biopsy; Procedure: Research blood sample

INTERVENTIONS:
Drug: Neratinib
  Other Names: PF-05208767
Drug: Fulvestrant
  Other Names: Faslodex
  Arms: Crossover: Neratinib + Fulvestrant + Trastuzumab; Part II: Neratinib + Fulvestrant (ER+, fulvestrant-naive); Part II: Neratinib + Fulvestrant (ER+. prior fulvestrant-tx)
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Crossover: Neratinib + Fulvestrant + Trastuzumab; Crossover: Neratinib + Trastuzumab
Procedure: Tumor biopsy — -Optional at baseline and disease progression
Procedure: Research blood sample — -Baseline, cycle 1 day 15, cycle 2 day 1, cycle 3 day 1, day 1 of each odd cycle, end of treatment (progression)

SUMMARY:
This phase II study will test cancer to see if it has a HER2 mutation and, if so, see how HER2 mutated cancer responds to treatment with neratinib.

DETAILED DESCRIPTION:
Overexpression of HER2 due to gene amplification is an established therapeutic target in breast cancer for which multiple HER2 targeted drugs are now available. However, the majority of breast cancers are without HER2 overexpression/non-amplified and not currently eligible to receive HER2 targeted drugs. Advances in tumor genome sequencing technology led to the identification of recurrent HER2 mutations (HER2mut) in approximately 2% of HER2 non-amplified primary breast cancers, and 3-5% of metastatic tumors. Importantly, tumor cells harboring HER2mut are sensitive to the anti-tumor effects of HER2-targeted agents in preclinical models, especially neratinib, a potent irreversible pan-HER inhibitor. However, neratinib monotherapy has demonstrated only modest single agent activity in HER2mut,, non-amplified metastatic breast cancer (MBC). Based on the hypothesis that the combination of neratinib and fulvestrant will be more effective than neratinib alone in ER+/HER2mut, non-amplified MBC the investigators conducted a single arm phase II study of neratinib plus fulvestrant with 2 cohorts, fulvestrant (FUL)-treated and FUL-naïve, for patients with ER+/HER2mut, non-amplified MBC to assess the anti-tumor effects of this combination. An exploratory ER-negative (ER-) HER2mut cohort was also included for the efficacy of neratinib monotherapy.

ELIGIBILITY:
Inclusion Criteria for Pre-registration (for patients with unknown HER2 mutation status to have tumor tissue screened centrally by Washington University GPS laboratory):

* Histologically or cytologically confirmed HER2-negative (0 or 1+ by IHC or non-amplified by FISH) breast cancer that is stage IV.
* Agree to provide archival tumor material for research
* There is no limitation on the number of prior lines of systemic therapy.
* Presence of measurable or non-measurable disease by RECIST 1.1 is acceptable, except to be eligible for the Part II fulvestrant-naive ER+ cohort, at least one measurable disease by RECIST 1.1 is required.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Adequate organ function as defined below within 8 weeks of pre-registration:

  * Serum creatinine ≤1.5 x ULN
  * Chil-Pugh class A if with liver disease
* Able to understand and willing to sign an IRB approved written informed consent document.

Note: HER2 mutation testing may be performed while the patient is receiving active systemic therapy for metastatic breast cancer so that the result can be used to determine eligibility for study drug therapy in the future.

Exclusion Criteria for Pre-registration:

* Testing for LVEF is not required for pre-registration, but patient must not have a recent LVEF < LLN or have symptoms of congestive heart failure.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Acute or currently active hepatic or biliary disease requiring antiviral therapy (with the exception of Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment).
* History of significant cardiac disease, cardiac risk factors, or uncontrolled arrhythmias.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest.

Inclusion Criteria for Registration (for patients initially pre-registered and with HER2 mutation identified by Washington University GPS laboratory)

* Tumor tissue tested positive for HER2 mutation. HER2 mutations detected by Guardant360 are also eligible.
* Agree to provide archival tumor material for research
* ECOG performance status ≤2
* Adequate organ function as defined below within 2 weeks of registration:

  * ANC ≥1.5 x 10^9/L
  * Platelet count ≥100 x 10^9/L
  * Serum creatinine ≤1.5 x ULN
  * Child-Pugh class A if with liver disease
* The patient must have completed radiation therapy and be at least 1 week from the last systemic chemotherapy administration, with adequate recovery of bone marrow and organ functions, before starting neratinib.
* Presence of disease progression on the most recent disease evaluation.
* Patients with known brain metastasis are eligible, but must have received radiation and be off steroids and stable (without evidence of disease progression by imaging or exam) for 3 months.
* QTc interval ≤450 msec for men or < or ≤ 470 msec for women within 2 weeks of registration.
* LVEF > or = institutional ILLN within 4 weeks of registration.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men must agree and commit to use a barrier method of contraception while on treatment and for 3 months after the last dose of the investigational product.
* Able to understand and willing to sign an IRB approved written informed consent document.
* There is no limitation on the number of prior lines of systemic therapy.
* To be eligible for the Part II fulvestrant-naive ER+ cohort, prior treatment with fulvestrant is not allowed. In addition, ER and/or PR positivity by institutional standard is required on pathology from the most recent tumor specimen if biopsy was done unless the tissue source (for example, pleural effusion or ascites or bone biopsy) may yield false negative ER and/or PR result, in which case the pathology from an earlier time point could be used and a discussion with the study chair is required.
* To be eligible for the Part II fulvestrant-treated ER+ cohort, prior disease progression on fulvestrant is required. In addition, ER and/or PR positivity by institutional standard is required on pathology from the most recent tumor specimen unless the tissue source (for example, pleural effusion or ascites or bone biopsy) may yield false negative ER and/or PR result, in which case the pathology form an earlier time point could be used and a discussion with the study chair is required.

Inclusion Criteria for Registration (for patients with HER2 mutation identified at an outside CLIA certified location):

* Histologically or cytologically confirmed HER2-negative (0 or 1+ by IHC or non-amplified by FISH) breast cancer that is stage IV.
* Tumor tissue or circulating tumor DNA tested positive for HER2 mutation. Mutations outside the list will be assessed on a case-by-case basis by the study team to determine eligibility.
* Presence of measurable or non-measurable disease by RECIST 1.1 is acceptable, except to be eligible for the Part II fulvestrant-naïve ER+ cohort, at least one measurable disease by RECIST 1.1 is required.
* At least 18 years of age.
* ECOG performance status < 2 (see Appendix A).
* Adequate organ function as defined below within 2 weeks of registration:

  * Absolute neutrophil count: ≥1.5 × 109/L (1500/mm3)
  * Platelet count: ≥100 × 109/L (100,000/mm3)
  * Serum creatinine: ≤1.5 x ULN
  * Child-Pugh class A if with liver disease
* The patient must have completed radiation therapy and be at least 1 week from the last systemic therapy administration, with adequate recovery of bone marrow and organ functions, before starting neratinib.
* Presence of disease progression on the most recent disease evaluation.
* Patients with known treated brain metastasis are eligible, but must have received radiation and be off steroids and stable (without evidence of disease progression by imaging or exam) for 3 months.
* QTc interval ≤ 450 msec for men or ≤ 470 msec for women within 2 weeks of registration.
* LVEF > institutional LLN within 4 weeks of registration.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men must agree and commit to use a barrier method of contraception while on treatment and for 3 months after the last dose of the investigational product
* Able to understand and willing to sign an IRB approved written informed consent document.
* There is no limitation on the number of prior lines of systemic therapy.
* To be eligible for the Part II fulvestrant-naïve ER+ cohort, prior treatment with fulvestrant is not allowed. In addition, ER and/or PR positivity by institutional standard is required on pathology from the most recent tumor specimen if biopsy was done unless the tissue source (for example, pleural effusion or ascites or bone biopsy) may yield false negative ER and/or PR result, in which case the pathology from an earlier time point could be used and a discussion with the study chair is required.
* To be eligible for the Part II fulvestrant-treated ER+ cohort, prior disease progression on fulvestrant is required. In addition, ER and/or PR positivity by institutional standard is required on pathology from the most recent tumor specimen unless the tissue source (for example, pleural effusion or ascites or bone biopsy) may yield false negative ER and/or PR result, in which case the pathology from an earlier time point could be used and a discussion with the study chair is required.

Exclusion Criteria for Registration:

* Currently receiving any other investigational agents or systemic cancer therapy.
* Currently taking medications and herbal or dietary supplements that are strong cytochrome P450 (CYP) 3A4 inducers or inhibitors. The washout period must have been completed prior to the start of neratinib if the patient was taking any of these agents. If unavoidable, patients taking CYP3A4 inhibitors should be monitored closely.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Acute or currently active/requiring antiviral therapy hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment).
* Pregnant and/or breastfeeding.
* History of significant cardiac disease, cardiac risk factors, or uncontrolled arrhythmias.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest.
* Experiencing grade 2 or greater diarrhea.
* Prior treatment with neratinib
* Child-Pugh class B or C liver dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, M.D., Ph.D, Principal Investigator — Washington University School of Medicine
Locations (17):
- United States (15):
  - University of Alabama Cancer Center, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - Stanford Medicine Cancer Institute, Stanford, California
  - University of Miami Hospital and Clinics, Miami, Florida
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Harvard University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina at Chapel Hill (Lineberger Comprehensive Cancer Center), Chapel Hill, North Carolina
  - Duke Cancer Institute at Duke University Medical Center, Durham, North Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jhaveri K, Eli LD, Wildiers H, Hurvitz SA, Guerrero-Zotano A, Unni N, Brufsky A, Park H, Waisman J, Yang ES, Spanggaard I, Reid S, Burkard ME, Vinayak S, Prat A, Arnedos M, Bidard FC, Loi S, Crown J, Bhave M, Piha-Paul SA, Suga JM, Chia S, Saura C, Garcia-Saenz JA, Gambardella V, de Miguel MJ, Gal-Yam EN, Rapael A, Stemmer SM, Ma C, Hanker AB, Ye D, Goldman JW, Bose R, Peterson L, Bell JSK, Frazier A, DiPrimeo D, Wong A, Arteaga CL, Solit DB. Neratinib + fulvestrant + trastuzumab for HR-positive, HER2-negative, HER2-mutant metastatic breast cancer: outcomes and biomarker analysis from the SUMMIT trial. Ann Oncol. 2023 Oct;34(10):885-898. doi: 10.1016/j.annonc.2023.08.003. Epub 2023 Aug 18. PMID 37597578
- [Derived] Shishido SN, Masson R, Xu L, Welter L, Prabakar RK, D' Souza A, Spicer D, Kang I, Jayachandran P, Hicks J, Lu J, Kuhn P. Disease characterization in liquid biopsy from HER2-mutated, non-amplified metastatic breast cancer patients treated with neratinib. NPJ Breast Cancer. 2022 Feb 18;8(1):22. doi: 10.1038/s41523-022-00390-5. PMID 35181666
- [Derived] Exman P, Garrido-Castro AC, Hughes ME, Freedman RA, Li T, Trippa L, Bychkovsky BL, Barroso-Sousa R, Di Lascio S, Mackichan C, Lloyd MR, Krevalin M, Cerami E, Merrill MS, Santiago R, Crowley L, Kuhnly N, Files J, Lindeman NI, MacConaill LE, Kumari P, Tolaney SM, Krop IE, Bose R, Johnson BE, Ma CX, Dillon DA, Winer EP, Wagle N, Lin NU. Identifying ERBB2 Activating Mutations in HER2-Negative Breast Cancer: Clinical Impact of Institute-Wide Genomic Testing and Enrollment in Matched Therapy Trials. JCO Precis Oncol. 2019 Nov 15;3:PO.19.00087. doi: 10.1200/PO.19.00087. eCollection 2019. PMID 32923853
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Part I and Part 2
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Started | 16 | 5 | 11 | 24 | 0 | 0
Completed | 16 | 4 | 10 | 21 | 0 | 0
Not Completed | 0 | 1 | 1 | 3 | 0 | 0
Not completed — Grade 2 vomiting and progressive disease | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Grade 3 diarrhea and withdrawal | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Grade 2 vomiting | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Grade 3 dizziness and progressive disease | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Grade 3 diarrhea and duodenal ulcer | 0 | 0 | 0 | 1 | 0 | 0
Period: Crossover
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Started | 0 | 0 | 0 | 0 | 3 | 5
Completed | 0 | 0 | 0 | 0 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Total
Number analyzed (Participants) | 16 | 5 | 11 | 24 | 56
Age, Continuous [Median (Full Range); unit: years] | 58 [31 to 74] | 63 [58 to 67] | 58 [41 to 82] | 64 [35 to 76] | 61 [31 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 10 | 24 | 55
  Male | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 16 | 5 | 9 | 17 | 47
  Unknown or Not Reported | 0 | 0 | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 5
  White | 13 | 4 | 8 | 23 | 48
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 0 | 0 | 0 | 0
  United States | 14 | 5 | 11 | 24 | 56
HER2 Status [Count of Participants; unit: Participants]
  Activating | 15 | 5 | 11 | 24 | 55
  Novel | 1 | 0 | 0 | 0 | 1
Histology Subtype [Count of Participants; unit: Participants]
  Ductal | 10 | 3 | 7 | 10 | 30
  Lobular | 5 | 2 | 2 | 12 | 21
  Other | 1 | 0 | 1 | 2 | 4
  Unknown | 0 | 0 | 1 | 0 | 1
Tumor Grade [Count of Participants; unit: Participants] — * Cancer cells are graded when they are removed from the breast. The grade is based on how much the cancer cells look like normal cells.
  * A low grade number (grade 1) usually means the cancer is slower-growing and less likely to spread.
  * An intermediate grade number (grade 2) means the cancer is growing faster than a grade 1 cancer but slower than a grade 3 cancer.
  * A high grade number (grade 3) means a faster-growing cancer that's more likely to spread.
  Participants
    I/II | 8 | 0 | 5 | 12 | 25
    II | 1 | 1 | 0 | 3 | 5
    III | 7 | 4 | 2 | 3 | 16
    Unknown | 0 | 0 | 4 | 6 | 10
Tumor Stage at Initial Diagnosis [Count of Participants; unit: Participants] — * Staging occurred at initial diagnosis after physical exam, mammogram, and other diagnostic imaging tests. The staging also takes into account pathology reports from the breast biopsy or surgery.
  * Stage I has a better outcome than Stage IV.
  Participants
    I | 2 | 1 | 2 | 4 | 9
    II | 6 | 2 | 3 | 9 | 20
    IIA | 0 | 0 | 1 | 0 | 1
    IIB | 2 | 0 | 0 | 0 | 2
    III | 4 | 1 | 0 | 4 | 9
    IIIA | 0 | 0 | 0 | 3 | 3
    IIIC | 0 | 0 | 0 | 1 | 1
    IV | 1 | 1 | 2 | 1 | 5
    Unknown | 1 | 0 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part I Only: Clinical Benefit Rate (CR+PR+SD≥6months) of Patients Who Received Neratinib Alone
Description: * Imaging for clinical benefit rate occurred at baseline (for an initial comparison scan) and every 2 cycles (28 day length) thereafter.
  * Complete response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have had stable disease for at least 6 months.
Time Frame: Through completion of treatment (median treatment time of 90 days, full range 54-716 days)
Population: Only Part I participants were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 16 | 0 | 0 | 0 | 0 | 0
Participants | 5 |  |  |  |  |

2. Primary Outcome: Part II ER-cohort Only: Clinical Benefit Rate (CR+PR+SD≥6months) of Neratinib in Patients With Metastatic HER2-, ER- Breast Cancer That Carry HER2 Mutation
Description: as for outcome 1
Time Frame: Through completion of treatment (median treatment time of 62 days, full range 56-413 days)
Population: Only participants enrolled in the Part II ER-cohort are evaluable for this outcome measure. One participant was not evaluable in this cohort as the participant stopped treatment in cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 4 | 0 | 0 | 0 | 0
Participants |  | 1 |  |  |  |

3. Primary Outcome: Part II Fulvestrant-naive ER+ Cohort Only: Clinical Benefit (CR+PR+SD≥6 Months) of Neratinib + Fulvestrant in Patients With Metastatic HER2- ER+ Fulvestrant-naive Breast Cancer That Carry HER2 Mutation
Description: as for outcome 1
Time Frame: Through completion of treatment (median treatment time of 140.5 days, full range 48-770 days)
Population: Only participants enrolled in the Part II fulvestrant-naive ER+ cohort is evaluable for this outcome measure. One participant was not evaluable in this cohort as the participant stopped treatment in cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 0 | 10 | 0 | 0 | 0
Participants |  |  | 3 |  |  |

4. Primary Outcome: Part II Fulvestrant-treated ER+ Cohort Only: Clinical Benefit Rate (CR+PR+SD≥6months) of Neratinib + Fulvestrant in Patients With Metastatic HER2- ER+ Fulvestrant-treated Breast Cancer That Carry HER2 Mutation
Description: as for outcome 1
Time Frame: Through completion of treatment (median treatment time of 168 days, full range 28-671 days)
Population: Only participants enrolled in the fulvestrant-treated ER+ cohort are evaluable for this outcome measure. Three participants were not evaluable in this cohort as the participants stopped treatment in cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 0 | 0 | 21 | 0 | 0
Participants |  |  |  | 8 |  |

5. Secondary Outcome: Progression-free Survival (PFS) of Patients Treated With Neratinib Alone in Patients With Metastatic HER2- But HER2 Mutated Breast Cancer by ER Status and by HER2 Mutations (Activating Versus Unknown Significance)
Description: * Participants were followed for progressive disease from start of treatment until completion of follow-up.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Through completion of follow-up; follow-up was through 30 days following completion of treatment (median follow-up of 92 days, full range 86 days-443 days)
Population: Only participants enrolled in the Part II ER-cohort are evaluable for this outcome measure. One participant was not evaluable in this cohort as the participant stopped treatment in cycle 1. The data represents exact number of weeks that each participant had progression-free survival. 2 participants with Activating mutation - S310F both had 8 weeks of PFS.
Measure: Number; unit: weeks
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 4 | 0 | 0 | 0 | 0
weeks
  Activating mutation - L7L755S: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Activating mutation - L7L755S |  | 9 |  |  |  |
  Activating mutation - S310F: number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0
  Activating mutation - S310F |  | 8 |  |  |  |
  Activating mutation - A775_G776insYVMA: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Activating mutation - A775_G776insYVMA |  | 17 |  |  |  |

6. Secondary Outcome: Number of Participants With HER2 Mutation Subtype and Histology Subtype
Time Frame: At the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx)
Number analyzed (Participants) | 16 | 5 | 11 | 24
Participants
  ECD mutation : Ductal histology | 3 | 1 | 1 | 1
  ECD mutation : Other histology | 0 | 1 | 1 | 2
  Exon 20 ins mutation : Ductal histology | 2 | 0 | 1 | 2
  Exon 20 ins mutation : Other histology | 2 | 1 | 0 | 2
  KD mutation : Ductal histology | 5 | 1 | 5 | 7
  KD mutation : Other histology | 4 | 1 | 3 | 10

7. Secondary Outcome: Number of Participants With HER2 Mutation Subtype and Tumor Grade
Description: -Cancer cells are graded when they are removed from the breast. The grade is based on how much the cancer cells look like normal cells.
  * A low grade number (grade 1) usually means the cancer is slower-growing and less likely to spread.
  * An intermediate grade number (grade 2) means the cancer is growing faster than a grade 1 cancer but slower than a grade 3 cancer.
  * A high grade number (grade 3) means a faster-growing cancer that's more likely to spread.
Time Frame: A time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx)
Number analyzed (Participants) | 16 | 5 | 11 | 24
Participants
  ECD mutation : Tumor grade I/II | 2 | 0 | 1 | 2
  ECD mutation : Tumor grade III | 1 | 3 | 0 | 0
  ECD mutation : Unknown | 0 | 0 | 1 | 1
  Exon 20 ins mutation : Tumor grade I/II | 1 | 1 | 0 | 2
  Exon 20 ins mutation : Tumor grade III | 3 | 0 | 1 | 0
  Exon 20 ins mutation : Unknown | 0 | 0 | 0 | 2
  KD mutation : Tumor grade I/II | 6 | 0 | 4 | 11
  KD mutation : Tumor grade III | 3 | 2 | 1 | 3
  KD mutation : Unknown | 0 | 0 | 3 | 3

8. Secondary Outcome: Correlate the Presence of HER2 Mutation Subtype With Tumor Staging at Initial Diagnosis
Description: * Staging occurred at initial diagnosis after physical exam, mammogram, and other diagnostic imaging tests. The staging also takes into account pathology reports from the breast biopsy or surgery.
  * Stage I has a better outcome than Stage IV.
Time Frame: At time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx)
Number analyzed (Participants) | 16 | 5 | 11 | 24
Participants
  ECD mutation : Stage I | 0 | 0 | 0 | 1
  ECD mutation : Stage II | 3 | 1 | 1 | 2
  ECD mutation : Stage III | 0 | 0 | 0 | 0
  ECD mutation : Stage IV | 0 | 1 | 0 | 0
  ECD mutation : Unknown | 0 | 0 | 1 | 0
  Exon 20 ins mutation : Stage I | 0 | 0 | 0 | 0
  Exon 20 ins mutation : Stage II | 3 | 0 | 1 | 1
  Exon 20 ins mutation : Stage III | 1 | 1 | 0 | 2
  Exon 20 ins mutation : Stage IV | 0 | 0 | 0 | 0
  Exon 20 ins mutation : Unknown | 0 | 0 | 0 | 1
  KD mutation : Stage I | 2 | 1 | 2 | 3
  KD mutation : Stage II | 2 | 1 | 2 | 6
  KD mutation : Stage III | 3 | 0 | 0 | 6
  KD mutation : Stage IV | 1 | 0 | 2 | 1
  KD mutation : Unknown | 1 | 0 | 2 | 1

9. Secondary Outcome: Correlate the Presence of HER2 Mutation Subtype With Progression-free Survival
Description: * Progression-free survival is defined as the number of weeks from start of treatment until disease progression or death.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Through completion of follow-up; follow-up was through 30 days following completion of treatment (median follow-up of 142 days, full range 54-800 days)
Population: The number analyzed for each row adds up to overall total number analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx)
Number analyzed (Participants) | 16 | 5 | 11 | 24
weeks
  ECD mutation: number analyzed (Participants) | 3 | 2 | 2 | 3
  ECD mutation | 11.0000 [9.0000 to 32.0000] | 8.0000 [NA to NA] — The sample size is too small to calculate the 95% confidence interval. | 48.5000 [16.0000 to 81.0000] | 3.0000 [1.0000 to 24.0000]
  Exon 20 ins mutation: number analyzed (Participants) | 4 | 1 | 1 | 4
  Exon 20 ins mutation | 26.0000 [8.0000 to 75.0000] | 17.0000 [NA to NA] — The sample size is too small to calculate the 95% confidence interval. | 26.000 [NA to NA] — The sample size is too small to calculate the 95% confidence interval. | 36.5000 [9.0000 to 68.0000]
  KD mutation: number analyzed (Participants) | 9 | 2 | 8 | 17
  KD mutation | 9.0000 [3.0000 to 31.0000] | 6.5000 [4.0000 to 9.0000] | 8.0000 [1.0000 to 24.0000] | 16.0000 [9.0000 to 27.0000]

10. Secondary Outcome: Part II ER-cohort Only: Progression-free Survival (PFS)
Description: as for outcome 9
Time Frame: Through completion of treatment (median treatment time of 62 days, full range 56-413 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 4 | 0 | 0 | 0 | 0
weeks |  | 8.5 [8 to NA] — There were too few participants with an event to calculate the upper limit of the confidence interval. |  |  |  |

11. Secondary Outcome: Part II Fulvestrant-naive ER+ Cohort Only: Progression-free Survival (PFS)
Description: as for outcome 9
Time Frame: Through completion of treatment (median treatment time of 140.5 days, full range 48-770 days)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 0 | 10 | 0 | 0 | 0
weeks |  |  | 20 [8 to NA] — There were too few participants with an event to calculate the upper limit of the confidence interval. |  |  |

12. Secondary Outcome: Part II Fulvestrant-treated ER+ Cohort Only: Progression-free Survival (PFS)
Description: as for outcome 9
Time Frame: Through completion of treatment (median treatment time of 168 days, full range 28-671 days)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 0 | 0 | 21 | 0 | 0
weeks |  |  |  | 24 [15.7 to 31] |  |

13. Secondary Outcome: Safety and Tolerability of Neratinib in Combination With Fulvestrant in Patients With HER2- ER+ HER2 Mutated Breast Cancer as Measured by Number of Participants With Related Adverse Events
Description: -CTCAE v 4.0 will be used to record adverse events. Related includes those possibly, probably, or definitely related to the treatment regimen.
Time Frame: Through completion of follow-up; follow-up was through 28 days following completion of treatment (median follow-up of 140 days, full range 52-798 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 16 | 5 | 11 | 24 | 3 | 5
Participants
  Anemia | 2 | 0 | 1 | 4 | 0 | 1
  LVEF Decrease | 0 | 0 | 0 | 0 | 1 | 0
  Heart failure with preserved ejection fraction | 0 | 0 | 0 | 0 | 0 | 1
  Tinnitus | 1 | 0 | 0 | 0 | 0 | 0
  Dry eye | 1 | 0 | 0 | 1 | 0 | 0
  Abdominal cramping | 1 | 0 | 0 | 0 | 0 | 0
  Abdominal pain | 0 | 0 | 2 | 3 | 0 | 0
  Bloating | 0 | 1 | 0 | 2 | 0 | 0
  Constipation | 5 | 0 | 1 | 2 | 0 | 0
  Diarrhea | 15 | 5 | 8 | 20 | 0 | 1
  Dry mouth | 0 | 0 | 0 | 4 | 0 | 0
  Dyspepsia | 2 | 0 | 1 | 6 | 0 | 0
  Flatulence | 0 | 0 | 0 | 1 | 0 | 0
  Mucositis oral | 3 | 0 | 0 | 2 | 0 | 0
  Nausea | 9 | 3 | 4 | 11 | 0 | 1
  Stomach pain | 1 | 0 | 0 | 0 | 0 | 0
  Stomatitis | 0 | 0 | 0 | 1 | 0 | 0
  Vomiting | 6 | 1 | 0 | 6 | 0 | 2
  Fatigue | 6 | 1 | 5 | 12 | 0 | 1
  Fever | 0 | 0 | 0 | 1 | 0 | 0
  Generalized weakness | 1 | 0 | 0 | 0 | 0 | 0
  Pain | 0 | 0 | 0 | 1 | 0 | 0
  Rhinitis infective | 0 | 0 | 0 | 1 | 0 | 0
  Upper respiratory infection | 0 | 0 | 0 | 1 | 0 | 0
  Urinary tract infection | 1 | 0 | 2 | 1 | 0 | 0
  Alaline aminotransferase increased | 3 | 0 | 2 | 4 | 0 | 1
  Alkaline phosphatase increased | 1 | 0 | 1 | 3 | 0 | 0
  Alkaline phosphatase decreased | 0 | 0 | 0 | 1 | 0 | 0
  Aspartate aminotransferase increased | 2 | 0 | 3 | 7 | 0 | 1
  CD4 lymphocytes decreased | 1 | 0 | 0 | 0 | 0 | 0
  Creatinine increased | 3 | 0 | 0 | 1 | 0 | 1
  Ejection fraction decreased | 0 | 0 | 0 | 0 | 1 | 0
  INR increased | 0 | 0 | 1 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 0 | 2 | 2 | 0 | 0
  Neutrophil count decreased | 0 | 0 | 0 | 2 | 0 | 1
  Platelet count decreased | 0 | 0 | 0 | 0 | 1 | 1
  Weight loss | 3 | 1 | 0 | 4 | 0 | 1
  White blood cell decreased | 0 | 0 | 0 | 4 | 0 | 0
  Anorexia | 7 | 1 | 7 | 9 | 0 | 2
  Dehydration | 3 | 1 | 1 | 6 | 1 | 1
  Hypercalcemia | 0 | 0 | 0 | 2 | 0 | 0
  Hyperglycemia | 1 | 0 | 0 | 2 | 0 | 0
  Hyperkalemia | 0 | 0 | 0 | 1 | 0 | 1
  Hypoalbuminemia | 2 | 0 | 0 | 1 | 0 | 0
  Hypocalcemia | 1 | 0 | 0 | 2 | 0 | 0
  Hypokalemia | 1 | 0 | 1 | 1 | 0 | 0
  Hyponatremia | 0 | 0 | 1 | 1 | 0 | 0
  Hypophosphatemia | 2 | 0 | 0 | 1 | 0 | 0
  Arthralgia | 1 | 0 | 0 | 2 | 0 | 0
  Back pain | 2 | 0 | 0 | 0 | 0 | 0
  Bone pain | 1 | 0 | 0 | 0 | 0 | 0
  Flank pain | 1 | 0 | 0 | 0 | 0 | 0
  Generalized muscle weakness | 0 | 0 | 0 | 2 | 0 | 0
  Joint range of motion decreased | 0 | 0 | 1 | 0 | 0 | 0
  Leg cramp | 1 | 0 | 0 | 0 | 0 | 0
  Muscle weakness left sided | 0 | 0 | 0 | 1 | 0 | 0
  Muscle weakness lower limb | 0 | 0 | 0 | 1 | 0 | 0
  Myalgia | 0 | 0 | 0 | 1 | 0 | 0
  Pain at injection site | 0 | 0 | 1 | 0 | 0 | 0
  Pain in extremity | 0 | 0 | 1 | 0 | 0 | 0
  Dizziness | 1 | 0 | 2 | 4 | 0 | 0
  Dysgeusia | 0 | 0 | 1 | 3 | 0 | 2
  Headache | 1 | 0 | 2 | 0 | 0 | 0
  Peripheral sensory neuropathy | 0 | 1 | 0 | 1 | 0 | 0
  Syncope | 1 | 0 | 1 | 0 | 0 | 0
  Depression | 0 | 0 | 1 | 0 | 0 | 0
  Insomnia | 0 | 0 | 1 | 0 | 0 | 0
  Acute kidney injury | 0 | 0 | 1 | 0 | 0 | 0
  Urinary tract obstruction | 0 | 0 | 1 | 0 | 0 | 0
  Urine discoloration | 0 | 0 | 1 | 1 | 0 | 0
  Urine odor | 0 | 0 | 1 | 0 | 0 | 0
  Cough | 1 | 0 | 0 | 1 | 0 | 0
  Dyspnea | 0 | 0 | 0 | 1 | 0 | 0
  Epistaxis | 0 | 0 | 1 | 0 | 0 | 0
  Hoarseness | 0 | 0 | 0 | 1 | 0 | 0
  Postnasal drip | 0 | 0 | 1 | 0 | 0 | 0
  Rhinorrhea | 0 | 0 | 0 | 1 | 0 | 0
  Alopecia | 1 | 0 | 0 | 0 | 0 | 0
  Dry hair | 1 | 0 | 0 | 0 | 0 | 0
  Dry skin | 0 | 0 | 0 | 2 | 0 | 0
  Nail changes | 1 | 0 | 0 | 1 | 0 | 0
  Pruritus | 1 | 0 | 0 | 1 | 0 | 1
  Rash acneiform | 0 | 0 | 2 | 4 | 0 | 0
  Rash maculopapular | 1 | 1 | 1 | 1 | 0 | 0
  Skin hyperpigmentation | 1 | 0 | 0 | 1 | 0 | 0
  Sterile abscess at subcutaneous injection site | 0 | 0 | 1 | 0 | 0 | 0
  Hot flashes | 1 | 0 | 1 | 1 | 0 | 0
  Hypotension | 1 | 0 | 1 | 1 | 0 | 0

14. Secondary Outcome: Part II Fulvestrant-naive ER+ Cohort Only: Response Rate (RR)
Description: * RR is defined as number of participants with complete response or partial response as best response.
  * Complete response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Through completion of treatment (median treatment time of 140.5 days, full range 48-770 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 0 | 10 | 0 | 0 | 0
Participants |  |  | 3 |  |  |

15. Secondary Outcome: Part II Fulvestrant-treated ER+ Cohort Only: Response Rate (RR)
Description: as for outcome 14
Time Frame: Through completion of treatment (median treatment time of 168 days, full range 28-671 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
Number analyzed (Participants) | 0 | 0 | 0 | 21 | 0 | 0
Participants |  |  |  | 5 |  |

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from start of treatment up to 28 days following the last day of study treatment. Median follow-up was 40 days, full range 52-798 days.
Arm/Group | Part I: Neratinib Only | Part II: Neratinib Only (ER-) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) | Crossover: Neratinib + Trastuzumab | Crossover: Neratinib + Fulvestrant + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 10/16 | 1/5 | 5/11 | 9/24 | 3/3 | 4/5
Serious Adverse Events (participants affected / at risk) | 5/16 | 1/5 | 2/11 | 9/24 | 2/3 | 0/5
Other Adverse Events (participants affected / at risk) | 16/16 | 5/5 | 11/11 | 24/24 | 3/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Neratinib Only (N=16) | Part II: Neratinib Only (ER-) (N=5) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) (N=11) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) (N=24) | Crossover: Neratinib + Trastuzumab (N=3) | Crossover: Neratinib + Fulvestrant + Trastuzumab (N=5)
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bell's palsy (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 2 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2 | 0 | 0
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Expressive aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: Neratinib Only (N=16) | Part II: Neratinib Only (ER-) (N=5) | Part II: Neratinib + Fulvestrant (ER+, Fulvestrant-naive) (N=11) | Part II: Neratinib + Fulvestrant (ER+. Prior Fulvestrant-tx) (N=24) | Crossover: Neratinib + Trastuzumab (N=3) | Crossover: Neratinib + Fulvestrant + Trastuzumab (N=5)
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 6 | 2 | 1
Thrombotic thrombocytopenia purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
LVEF decrease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0
Blurred vision (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Double vision (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Itchy eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral vision change (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Styes (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Abdominal cramping (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Abdominal fullness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 5 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 9 | 1 | 3 | 9 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 16 | 5 | 9 | 22 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 6 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal illness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 4 | 4 | 12 | 0 | 2
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 10 | 1 | 1 | 6 | 0 | 3
Changes in dentition (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 1 | 2 | 2 | 0
Failure-to-thrive (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 0 | 5 | 12 | 0 | 1
Fever (General disorders) | 0 | 0 | 2 | 5 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Generalized weakness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 2 | 1 | 0
Pain (General disorders) | 4 | 0 | 0 | 3 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bilateral breast infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cold (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gum infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Shingles (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Stomach bug (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Strep throat (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 3 | 4 | 1 | 2
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1
Finger pad cut off (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 3 | 5 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1 | 2 | 6 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 5 | 8 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 3 | 0 | 0 | 2 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 1 | 2 | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 2 | 0 | 1
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0 | 1 | 1
Weight loss (Investigations) | 5 | 1 | 0 | 4 | 1 | 2
White blood cell decreased (Investigations) | 0 | 0 | 0 | 4 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 10 | 1 | 7 | 10 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 1 | 5 | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 3 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 5 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 1 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 2 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1 | 0 | 0
Hypoproteinemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Type 2 Diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 4 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 0 | 1
Finger pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 0 | 0
Gait disturbance (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leg cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Pain at injection site (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0 | 0
Shoulder tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
New brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 5 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 3 | 0 | 2
Expressive aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 2 | 2 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Altered mental status (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 1 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 0 | 1 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bilateral ureteral stent placement (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Urine odor (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 4 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 6 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Nose irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Bug bite (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry hair (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
New skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 4 | 0 | 0
Rash maculopapular (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Sterile abscess at subcutaneous injection site (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bilateral percutaneous nephrostomy tubes placement (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Chest wall port placement (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Nephrostomy tubes exchange (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 2 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 2 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT01670877/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT01670877/ICF_001.pdf